CLINICAL TRIAL: NCT00514592
Title: Additional Neurological Symptoms Before Surgery of the Carotid Arteries - A Prospective Study
Brief Title: Additional Neurological Symptoms Before Surgery of the Carotid Arteries - A Prospective Study (ANSYSCAP)
Acronym: ANSYSCAP
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Elias Johansson, MD, PhD, Umeå University
Other Study IDs: EJ-0418
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-09

CONDITIONS: Carotid Stenoses
Keywords: Carotid stenosis; Carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: All patients enter the same group
  Interventions: Other: New Guidelines

INTERVENTIONS:
Other: New Guidelines — New practical guidelines after half of the study aimed at reducing the delay and increasing the patient safety.

SUMMARY:
A single center observational study. Observing the time between cerebrovascular symptoms and Carotid Endarterectomy (CEA) and patient outcome. An intervention at 17 of the 29 study months aimed at reducing the delay and increasing the patient safety. Main outcome is to measure the reduction in recurrent stroke with decreased delay to CEA.

DETAILED DESCRIPTION:
All patients with a carotid stenosis >50% according to the NASCET-criteria are included. The study does not affect the health care the patients receive. The time between symptom and surgery is compared to the outcome of the CEA after 45 days, 6 months, 1 year and 5 years. An intervention in the form of new practical local and regional guidelines in January 2009 (#17 of the 29 study months) aimed at reducing the delay and increasing the patient safety.

PRIMARY AIM:

To study the risk of Ipsilateral stroke, any stroke, death, any cerebrovascular event, any cardiovascular event.

Two primary analyses:

1. Ipsilateral ischemic stroke within 90 Days of the presenting event. This analysis is aimed at the short term risk of pre-operative stroke. Survival analysis will be used. CEA will be used a censor, thus excluding all peri-operative and postoperative strokes.
2. All primary endpoints within 5 years of the presenting event. This analysis is aimed att the long term risk of cardio-vascular morbidity and mortality.

Secondary analyses:

1) Same as first primary analysis, but including all stroke as endpoint, not only ipsilateral ischemic stroke.

SECONDARY AIM:

To attempt to validate different risk and score systems already published by other sources. Such as can ABCD2-score be used safely to chose between acute and fast normal screening for carotid stenosis?

ELIGIBILITY:
Inclusion Criteria:

* Carotid stenosis >50% according to NASCET criteria

Exclusion Criteria:

* Not preliminary judged as having an indication for surgery, before an extensive investigation is launched. Thus, some patients that will not undergo CEA will be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a carotid stenosis >50%, preliminary eligable for CEA in the northern region of Sweden
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per G Wester, Prof., Principal Investigator
Locations (1):
- University Hospital, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Rothwell PM, Eliasziw M, Gutnikov SA, Warlow CP, Barnett HJ; Carotid Endarterectomy Trialists Collaboration. Endarterectomy for symptomatic carotid stenosis in relation to clinical subgroups and timing of surgery. Lancet. 2004 Mar 20;363(9413):915-24. doi: 10.1016/S0140-6736(04)15785-1. PMID 15043958

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients enter the same group
Period: Overall Study
Arm/Group | All Patients
Started | 230
Completed | 230
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients are in the same group
Arm/Group | All Patients
Number analyzed (Participants) | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 147

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Ischemic Stroke Before Carotid Endarterectomy
Description: Ipsilateral ischemic stroke after the presenting event. Only events that occurs within 90 days and before Carotid EndArterectomy (CEA) is used.
Time Frame: Before CEA
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 230
participants | 33

2. Secondary Outcome: Any Stroke Before Carotid Enderarterectomy
Description: Same as primary endpoint, but includes stroke of all types.
Time Frame: Before CEA
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 230
participants | 36

ADVERSE EVENTS:
Time Frame: Adverse events not recorded other than the primary and secodary endpoint.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/230
Other Adverse Events (participants affected / at risk) | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes